CLINICAL TRIAL: NCT05732467
Title: Effectiveness of Virtual Reality Training in Amblyopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0755
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Amblyopia
Keywords: amblyopia; virtual reality
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Device: visual function training software; Other: corrective glasses
- control group (Other)
  Interventions: Other: occlusion therapy; Other: corrective glasses

INTERVENTIONS:
Device: visual function training software — Experimental group: If there is a refractive problem, first correct the refraction, wear corrective glasses, and then use visual function training therapy software (model: SJ-JRS2021) for treatment.
  Other Names: visual function training software (model: SJ-JRS2021)
  Arms: experimental group
Other: occlusion therapy — Control group: If there is a refractive problem, correct the refraction first, wear corrective glasses combined with occlusion therapy, and cover the fellow eye for 2 hours a day.
  Arms: control group
Other: corrective glasses — corrective glasses

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of visual function training software (model: SJ-JRS2021) in the treatment of mild to moderate amblyopia in children. The main questions it aims to answer are:

* Whether virtual reality training is more effective than occlusion therapy
* Safety of virtual reality training in amblyopia treatment If participants have refractive problems, correct the refraction first and wear corrective glasses. The experimental group will be treated using visual function training therapy software (model: SJ-JRS2021). The control group will be treated with occlusion therapy covering the contralateral eye for 2 hours a day. Researchers will compare experimental group with control group to see if the experimental group has better corrected vision recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-7 years old (including 4 and 7 years old), both sexes;
* Monocular amblyopia was diagnosed;
* The corrected visual acuity of amblyopia is between 0.2 (inclusive) and 0.6, and the binocular visual difference is more than 2 lines;
* The guardian of the subject can understand the purpose of the trial and sign the informed consent. The subject can cooperate with the treatment and related ophthalmic examination

Exclusion Criteria:

* The subject has tumor, heart disease, hypertension and epilepsy;
* The subject has an implanted electronic device, such as a pacemaker;
* The subject has suffered from mental illness;
* Subject suffers from vertigo, fear of heights or brain trauma;
* The subject has photophobia and tears caused by keratitis, conjunctivitis, internal trichiasis and other diseases at any time;
* The subject has strabismus or congenital cataract, congenital ptosis, trauma and other ocular organic lesions and related surgical history;
* Subject has had any form of treatment for amblyopia other than refractive correction and covering treatment.
* Other conditions, such as severe heart, liver and kidney disease, under which the investigator considers that the patient should not participate in the trial for safety reasons or in the interest of the patient.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | 16 weeks

SECONDARY OUTCOMES:
Near stereopsis | 16 weeks
contrast sensitivity | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiajing Tang, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China